CLINICAL TRIAL: NCT04428489
Title: A Follow-up Observational Study of ICUS and CCUS Patients
Brief Title: Follow-up Study of ICUS and CCUS Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Associate Professor, The First Affiliated Hospital of Soochow University
Other Study IDs: SZcytopenia01
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes
Keywords: Idiopathic cytopenia of undetermined significance (ICUS); Clonal cytopenia of unknown significance (CCUS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic cytopenia of undetermined significance (ICUS)
  Interventions: Other: Observation and necessary supportive care
- Clonal cytopenia of unknown significance (CCUS)
  Interventions: Other: Observation and necessary supportive care

INTERVENTIONS:
Other: Observation and necessary supportive care — For patients with ICUS and CCUS, necessary supportive care could be given. No addtitional treatment is administrated.

SUMMARY:
The proposed minimal diagnostic criteria for myelodysplastic syndromes (MDS) and potential pre-MDS conditions has been released by an international consensus group. Based on the criteria, patients with persistent cytopenia could be diagnosed with MDS, CCUS and ICUS. However, the process and outcome of pre-MDS conditions (CCUS, ICUS) is still to be characterized in Chinese population. We design this prospective observational study to explore the disease process and outcome in ICUS and CCUS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytopenia of any degree in one or more lineages: erythrocytes, neutrophils, or platelets. And the cytopenia has to be persistent (≥ 4 months) and lacking minimal diagnostic criteria of MDS.

Exclusion Criteria:

* Patients with cytopenia which could be explained by any other hematologic or non-hematologic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ICUS and CCUS based on the proposed minimal diagnostic criteria for myelodysplastic syndromes (MDS) and potential pre-MDS conditions
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Culumative transformation rate | 5 years
  Transformation is defined as progression from ICUS to CCUS, ICUS to MDS or CCUS to MDS. All patients are followed-up since entry into this trial and transformation events are recorded. Cumulative transformation rate is defined for all patients and estimated by competing risk methods.

SECONDARY OUTCOMES:
Event-free survival | 5 years
  Defined for all patients entry into this trial; measured from the date of entry into this trial to the date of progression or death from any cause; patients not known to have any of these events are censored on the date they were last examined.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided